CLINICAL TRIAL: NCT07075900
Title: Comparison of Effects of Dynamic Neuromuscular Stabilization Training and Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence: A Randomized Controlled Trial
Brief Title: Dynamic Neuromuscular Stabilization vs Pelvic Floor Muscle Training in Women With Stress Urinary Incontinence
Acronym: DYNA-SUI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Sevtap Günay, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DYNAPELVIS-SUI2025
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Stress Urinary Incontinence (SUI); Dynamic Neuromuscular Stabilization; Pelvic Floor Muscle Training; Muscle Morphology; Urinary Symptoms; Quality of Life
Keywords: stress urinary incontinence; dynamic neuromuscular stabilization; pelvic floor muscle training; physical activity; quality of life; muscle morphology
MeSH Terms: conditions — Urinary Incontinence, Stress; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DNS group (Experimental): Women aged 18-65 who have stress or stress-dominant mixed urinary incontinence. They are followed up for 12 weeks, consisting of 2 days/week face-to-face training sessions with the physiotherapist and 5 days/week sessions conducted by themselves.
  Interventions: Other: Dynamic Neuromuscular Stabilization Training
- PFMT group (Active Comparator): Women aged 18-65 who have stress or stress-dominant mixed urinary incontinence. They are followed up for 12 weeks, consisting of 2 days/week face-to-face training sessions with the physiotherapist and 5 days/week sessions conducted by themselves.
  Interventions: Other: Pelvic Floor Muscle Training
- Control (No Intervention): Receiving patient education only and no exercise was applied to the subjects included in the control group.

INTERVENTIONS:
Other: Dynamic Neuromuscular Stabilization Training — According to the principles of Dynamic Neuromuscular Stabilization (DNS), proper activation of the integrated spinal stabilization system requires that the abdominal muscles expand not only in the caudal direction but also posteriorly and laterally.Therefore, firstly, the physiotherapist will assess the expansion of the entire abdominal wall and teach the patient to regulate intra-abdominal pressure through correct breathing techniques. During training and exercises, a belt will be used. Participants will be instructed to maintain abdominal expansion toward the belt during exercises performed in positions supported by proper alignment. A four-phase exercise protocol based on developmental kinesiology principles will be implemented for the DNS group, beginning with supine-position exercises appropriate for the 3-month developmental stage.
  They will be instructed to repeat the exercises at least three times per day.Patients will record their home exercise program using an exercise diary.
  Arms: DNS group
Other: Pelvic Floor Muscle Training — Participants in the PFMT group will undergo a structured pelvic floor muscle training program supervised by a physiotherapist. The training will include verbal and manual instructions to ensure correct identification and isolated activation of the pelvic floor muscles without compensatory movements from the gluteal, abdominal, or thigh muscles using a NeuroTrac Simplex EMG-Biofeedback device.
  The exercise protocol will consist of both slow and fast contractions, focusing on endurance, strength, and coordination.
  The exercises will be performed in various positions (e.g., supine, sitting, standing) and will gradually progress in intensity and complexity over time, following the principles of motor learning stages. They will be instructed to repeat the exercises at least three times per day. Patients will record their home exercise program using an exercise diary.
  Arms: PFMT group

SUMMARY:
This randomized controlled trial aims to compare the pre- and post-treatment effects of Dynamic Neuromuscular Stabilization (DNS) training and Pelvic Floor Muscle Training (PFMT) on pelvic floor muscle function, pelvic floor morphometry, urinary symptoms, quality of life, sexual function, and physical activity levels in women with stress urinary incontinence (SUI).

Participants diagnosed with SUI by a specialist physician will be randomly assigned to one of three groups: DNS, PFMT, or a control group. Both DNS and PFMT interventions will be delivered as 12-week home exercise programs, performed five days a week and at least three times per day. To support adherence, participants will use an exercise diary. In addition, participants in the DNS and PFMT groups will attend the clinic twice a week for supervised sessions led by a physiotherapist.

The control group will receive a brochure containing lifestyle and bladder health recommendations but will not engage in any structured exercise program.

DETAILED DESCRIPTION:
Stress urinary incontinence (SUI) is defined by the International Continence Society as involuntary urine leakage due to insufficient urethral closure pressure during episodes of increased intra-abdominal pressure (IAP), such as coughing, sneezing, laughing, or physical activity. The continence mechanism involves intrinsic urethral closure, structural support of the urethra, and lumbopelvic stability. These components are interconnected through the endopelvic fascia and neural pathways.

The core musculature-including the diaphragm, transversus abdominis (TrA), pelvic floor muscles, and lumbar multifidus-functions synergistically within the myofascial system to regulate IAP. This coordination is essential for maintaining the optimal function of genitourinary organs, especially the bladder.

Dynamic Neuromuscular Stabilization (DNS) targets this integrated spinal stabilization system. DNS exercises are based on developmental kinesiology principles, comparing adult stabilization patterns to those of healthy infants. The goal is to retrain the neuromuscular system through repetitive, functional movements to restore automatic IAP regulation and trunk stability.

Although DNS has demonstrated clinical effectiveness in managing musculoskeletal disorders, cerebral palsy, hemiplegia, and athletic injuries, its role in the management of SUI remains underexplored. By promoting synchronous activation of the deep stabilizers-including the diaphragm, TrA, multifidus, and pelvic floor-DNS may offer a more comprehensive therapeutic approach than isolated pelvic floor muscle training.

In this context, the main questions of this study it aims to answer are:

Does Dynamic Neuromuscular Stabilization (DNS) training have an effect on pelvic floor muscle function, pelvic floor morphometry, symptoms, quality of life, sexual function, and physical activity levels in women with stress urinary incontinence (SUI)? Does Pelvic Floor Muscle Training (PFMT) improve pelvic floor muscle function, pelvic floor morphometry, symptoms, quality of life, sexual function, and physical activity levels in women with stress urinary incontinence (SUI)? Is there a difference between DNS exercises and PFMT in terms of their effects on pelvic floor muscle function, pelvic floor morphometry, symptoms, quality of life, sexual function, and physical activity levels before and after treatment in women with SUI?

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 65 years
* Diagnosed with stress urinary incontinence or stress-dominant mixed urinary incontinence by a specialist physician
* Having the ability to voluntarily contract the pelvic floor muscles
* Literate in Turkish
* Willing and voluntarily consenting to participate in the study

Exclusion Criteria:

* Pregnancy
* Presence of urgency-predominant urinary incontinence symptoms or fecal incontinence
* Inability to understand or cooperate with assessment procedures
* Presence of any neurological or rheumatological disease
* Severe cardiac or pulmonary disease
* Uncontrolled diabetes mellitus or hypertension
* Chronic liver and/or kidney failure
* Advanced pelvic organ prolapse (greater than grade 2)
* History of abdominal or pelvic surgery (including cesarean section) within the past year
* History of spinal surgery
* Current urinary tract infection
* History of pelvic radiation therapy
* Presence of spinal deformity
* History of acute low back pain within the past 4-6 weeks
* Receiving pelvic floor muscle training within the past three months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2025-07-16 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-Hour Pad test | Baseline and 12th week (at the end of the exercise program)
  The 1-hour pad test is a standardized objective measurement of urinary leakage under controlled physical activity conditions (e.g., walking, coughing, stair climbing). Participants wear a pre-weighed pad during the test; an increase in weight reflects urine loss. It is used to quantify the severity of stress urinary incontinence (SUI).
  Assessment Method: Pad weight difference in grams
Pelvic Floor Morphometry | Baseline and 12th week (at the end of the exercise program)
  3D transperineal ultrasonography allows objective morphometric and functional assessment of all compartments of the pelvic floor. 3D images are taken during rest, maximal voluntary contraction, and Valsalva maneuver, and measurements are recorded for levator ani muscle thickness, levator ani diameter, hiatal area, and the distance between the levator ani, urethra, and symphysis pubis. These measurements will be performed by a urogynecologist.
Pelvic Floor Muscle Strength and Endurance | Baseline and 12th week (at the end of the exercise program)
  The NeuroTract Simplex EMG-Biofeedback device will be used to assess pelvic floor muscle contraction strength (maximum squeeze pressure in cmH₂O or mmHg) and endurance (duration of sustained contraction). This provides an objective measure of muscle performance and training effect.
Incontinence Quality of Life Questionnaire (I-QOL) | Baseline and 12th week (at the end of the exercise program)
  The Incontinence Quality of Life Questionnaire (I-QOL) is a validated self-administered instrument that assesses the impact of urinary incontinence on quality of life a 22 items, including social embarrassment, avoidance behaviors, and psychosocial effects. Higher scores indicate a better perceived quality of life.
  A 2.5-point change in the I-QOL scale was determined to be the minimum clinically important difference (MCID) for women with urinary incontinence, representing a threshold at which patients typically report a noticeable improvement in quality of life. A 6.3-point improvement was predicted for the pre- and post-treatment assessment of the same group of women.
Incontinence Episodes and Number of Pads Used (from 3-Day Bladder Diary) | Baseline and 12th week (at the end of the exercise program)
  The number of incontinence episodes and the number of pads used are recorded by participants over three consecutive days. This provides a semi-objective reflection of symptom frequency and the daily impact of SUI.
  Assessment Tool: 3-Day Bladder Diary

SECONDARY OUTCOMES:
24-h Pad Test | Baseline and 12th week (at the end of the exercise program)
  A longer-duration objective measurement of urinary leakage. Participants wear a pre-weighed pad for 24 hours during typical daily activities. The post-use weight quantifies real-life incontinence severity.
  Assessment Method: Pad weight difference in grams
Frequency, Nocturia, and Fluid Intake | Baseline and 12th week (at the end of the exercise program)
  Additional parameters recorded in the bladder diary include daily voiding frequency, number of nocturnal voids (nocturia), and total fluid intake. These measures reflect bladder behavior and potential treatment-related improvements.
  Assessment Tool: 3-Day Bladder Diary
Pelvic Floor Muscle Strength (Digital Vaginal Palpation - Oxford Scale) | Baseline and 12th week (at the end of the exercise program)
  A trained physiotherapist will assess voluntary pelvic floor contractions using the Modified Oxford Scale (0= no contraction; 1= very weak; 2= weak; 3= moderate (with lifting); 4= good (with lifting); 5= strong (with lifting)). This semi-subjective but clinically accepted method provides a rapid evaluation of muscle activation ability.
  Assessment Method: Vaginal digital palpation
Female Sexual Function Index (FSFI) | Baseline and 12th week (at the end of the exercise program)
  A 19-item questionnaire evaluating six domains of female sexual function: desire, arousal, lubrication, orgasm, satisfaction, and pain. It is widely used in pelvic floor research and helps assess the broader quality-of-life effects of interventions.
  Scoring Range: 2-36 (higher scores = better function)
Physical Activity Levels | Baseline and 12th week (at the end of the exercise program)
  A validated questionnaire that quantifies physical activity levels across walking, moderate, and vigorous activities. Results are expressed in MET-minutes per week and allow for analysis of whether interventions affect physical activity engagement. The questionnaire consists of four separate sections and seven questions. It includes questions about the frequency of walking, moderate, and vigorous activities in the past week, and the time spent in these activities. The final question asks about the time spent sitting daily. Higher scores indicate a better outcome. According to the IPAQ scoring protocol, participants are classified into three categories based on total MET-minutes/week: Inactive (<600 MET-minutes/week ), Minimally Active (600-3000 MET-minutes/week ), and Health-Enhancing Physically Active (≥ 3000 MET-minutes/week) Assessment Tool: International Physical Activity Questionnaire - Short Form (IPAQ-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Kardelen ACAR, MSc, Principal Investigator — Izmir Katıp Celebi University, Institute of Health Sciences; Sevtap GUNAY UCURUM, Associate Professor, Study Director — Izmir Katıp Celebi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation; Ahmet Ozgur YENIEL, Professor, Study Chair — Ege University, Faculty of Medicine, Department of Obstetrics & Gynecology
Locations (1):
- Ege University, Faculty of Medicine, Department of Obstetrics & Gynecology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No